CLINICAL TRIAL: NCT00811772
Title: Comparison of the Long-term Effects on Mortality and Cardiovascular Morbidity of Percutaneous Coronary Intervention With Drug-eluting Stent Versus Bare-metal Stent. Randomized, Five-year Prospective, Multicenter Clinical Trial
Brief Title: Trial of Drug Eluting Stent Versus Bare Metal Stent to Treat Coronary Artery Stenosis
Acronym: NORSTENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Research Council of Norway (Other); The Royal Norwegian Ministry of Health (Other); Norwegian Council on Cardiovascular diseases (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 184916/V50 Res. council Norway; NSD19480; PREKNORD40/2008
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Coronary Atherosclerosis; Angina Pectoris; Myocardial Infarction
Keywords: Randomized controlled trial; Bare metal stent; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bare metal stent (Active Comparator): Implantation of one or more bare metal stent(s) to to treat coronary artery stenosis
  Interventions: Device: Percutaneous coronary intervention (PCI)
- Drug eluting stent (Experimental): Implantation of one or more drug eluting stent(s) to treat coronary artery stenosis
  Interventions: Device: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — Implantation of one or more bare metal stent(s)
  Arms: Bare metal stent
Device: Percutaneous coronary intervention (PCI) — Implantation of one or more drug eluting stent(s)
  Arms: Drug eluting stent

SUMMARY:
Stenosis of the coronary arteries may be treated by balloon dilatation followed by the implantation of a metal stent. However, restenosis occurs in 10-20% of patients treated with bare metal stents (BMS). Restenosis and treatment of restenosis is associated with risk of myocardial infarction (MI) and death. Drug eluting stents (DES)release drugs to the vessel wall that delay or inhibit the process of restenosis. Some reports have found that DES are associated with risk of acute stent thrombosis, MI and death. The precise magnitude of this risk is not known. Current evidence is therefore insufficient to balance the long-term risk and benefit of BMS vs DES.

The purpose of this trial is to compare the long-term effects on MI and total mortality of BMS vs DES. The trial will recruit 8000 patients from 8 Norwegian hospitals. The patients will be randomized to treatment with BMS or DES. Clinical events will be registered for 5 years after treatment. The study hypothesis is that there is no difference in the risk of death or myocardial infarction after treatment with BMS vs DES. The trial is initiated and run by university researchers and is sponsored by not-for-profit organizations.

DETAILED DESCRIPTION:
Background:

The balance of the long-term risks and benefits of coronary drug-eluting stents versus bare metal stents is not known.

Study objective:

The primary objective of the trial is to compare in a real-world setting the long-term effects on the incidence of death and myocardial infarction (composite primary end-point) after implantation of drug-eluting stents versus bare-metal stents. The secondary objective is to compare the long-term effects on the incidence of total death, cardiovascular deaths, major cardiovascular events, angina pectoris, revascularization procedures, and on health-related quality of life after implantation of drug-eluting stents versus bare-metal stents. The main tertiary objective is to assess the safety and efficacy in patient subgroups with specific demographic, clinical, and vessel- or lesion characteristics, and to conduct a cost-effectiveness analysis.

Study design:

This is a randomized, five-year prospective, multicenter, open-label clinical trial with blinded end point-evaluation.

Setting:

Investigator initiated trial conducted at 8 Norwegian interventional centres. The trial is sponsored by the Norwegian Research Council, the Regional Health Authorities and other not-for-profit organizations.

Randomization:

Patients will be randomized to receive either drug-eluting stent(s) or a bare-metal stent(s) in a 1:1 ratio.

Patients:

The trial will include 9000 patients with de novo lesions in native coronary arteries or by-pass grafts who meet the eligibility criteria. Men and women with stable angina pectoris or acute coronary syndrome will be included.

End-point:

The primary composite end point is total death and nonfatal myocardial infarction.Secondary end-points include total death and subcategories of death, fatal and nonfatal myocardial infarction, fatal and nonfatal stroke, angina pectoris, revascularization, major bleeding, health-related quality of life.

Length of follow-up:

Five years.

End-points collected by electronic linkage to national registries:

The trial will use the unique Norwegian 11-digit person number to search the National Patient Registry and the National Death Registry for nonfatal and fatal end-points during follow-up, thereby minimizing loss to follow-up. Information on angina pectoris and health-related quality of life will be collected by questionnaires.

Statistical power:

The trial has a statistical power of 93 percent to detect a three percent (RR 1.176) absolute difference in incidence between the study groups, and a power of 64 percent to detect a two percent (RR 1.118) absolute difference, given a two-sided alpha value of 0.05.

Statistical analysis:

Statistical analyses will be conducted according to the intention-to-treat principle, and will be performed by using widely accepted statistical and/or graphical software.

Data collection:

Electronic Case Record Form (e-CRF)

Clinical Event Committee:

Adjudication of all end-points according to pre-specified and standardized criteria by Clinical Event Committee blinded to study assignment.

Expected Timelines:

First patient enrollment: September 2008 Last patient enrollment: February 2011 Completion of Follow-up: December 2014.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >18 years with stable angina pectoris or acute coronary syndrome
* The patient has consented to participate and has signed the patient informed consent form
* All lesions requiring intervention in one or more native coronary artery/coronary artery by-pass graft are amendable for implantation of drug-eluting stents only, or bare-metal stents only.
* The patient has a unique 11-digit Norwegian person number, is able to communicate in Norwegian, and is expected not to emigrate during study follow-up.

Exclusion Criteria:

* Previous implantation of a coronary bare metal stent or coronary drug eluting stent
* Planned intervention of a bifurcation lesion with overlapping 2-stent technique
* The patient has a serious medical condition (other than coronary artery disease) with a life expectancy less than 5 years
* The patient is currently participating in another randomized trial that clinically interferes with the present trial, or requires coronary angiography or other coronary artery imaging procedures
* Hypersensitivity or allergies to drugs or components in use with percutaneous coronary intervention
* Contraindications for treatment with clopidogrel/ticlid for 9-12 months
* Patient is receiving chronic anticoagulation therapy (e.g., warfarin, heparin)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9013 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
First occurrence of all-cause mortality and non-fatal myocardial infarction (composite) | After five years of follow-up

SECONDARY OUTCOMES:
Major cardiovascular events | After five years of follow-up
Health related quality of life | After 6 months and then yearly for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kaare H Bønaa, MD, PhD, Principal Investigator — Dept of Heart Disease, St.Olavs University Hospital, Trondheim, Norway; Norwegian University of Science and Technology, Trondheim, Norway; University of Tromsø, Tromsø, Norway; Jan E Nordrehaug, MD, PhD, Study Chair — Department of Heart Disease, Haukeland University Hospital, Bergen, and University of Bergen, Bergen, Norway
Locations (8):
- Norway (8):
  - Department of Medicine, Sørlandet sykehus Arendal, Arendal
  - Department of Heart Disease, Haukeland University Hospital, Bergen
  - Department of Heart Disease, Feiringklinikken AS, Feiring
  - Department of Heart Disease, Rikshospitalet HF, Oslo
  - Department of Heart and Vascular Radiology and Department of Heart Disease, Ullevål University Hospital, Oslo
  - Department of Heart Disease, Stavanger University Hospital, Stavanger
  - Department of Heart Disease, University Hospital of Northern Norway, Tromsø
  - Department of Heart Disease, St.Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nordrehaug JE, Wiseth R, Bonaa KH. Drug-Eluting or Bare-Metal Stents for Coronary Artery Disease. N Engl J Med. 2016 Dec 29;375(26):2604-2605. doi: 10.1056/NEJMc1613866. No abstract available. PMID 28029911
- [Result] Bonaa KH, Mannsverk J, Wiseth R, Aaberge L, Myreng Y, Nygard O, Nilsen DW, Klow NE, Uchto M, Trovik T, Bendz B, Stavnes S, Bjornerheim R, Larsen AI, Slette M, Steigen T, Jakobsen OJ, Bleie O, Fossum E, Hanssen TA, Dahl-Eriksen O, Njolstad I, Rasmussen K, Wilsgaard T, Nordrehaug JE; NORSTENT Investigators. Drug-Eluting or Bare-Metal Stents for Coronary Artery Disease. N Engl J Med. 2016 Sep 29;375(13):1242-52. doi: 10.1056/NEJMoa1607991. Epub 2016 Aug 29. PMID 27572953
- [Derived] Samuelsen PJ, Eggen AE, Steigen T, Wilsgaard T, Kristensen A, Skogsholm A, Holme E, van den Heuvel C, Nordrehaug JE, Bendz B, Nilsen DWT, Bonaa KH. Incidence and risk factors for major bleeding among patients undergoing percutaneous coronary intervention: Findings from the Norwegian Coronary Stent Trial (NORSTENT). PLoS One. 2021 Mar 4;16(3):e0247358. doi: 10.1371/journal.pone.0247358. eCollection 2021. PMID 33661918